CLINICAL TRIAL: NCT05737524
Title: Virtually Assisted Home Rehabilitation After Acute Stroke-2 (VAST-rehab2)
Brief Title: Virtually Assisted Home Rehabilitation After Acute Stroke-2
Acronym: (VAST-rehab2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Lone Star Stroke Consortium (Unknown)
Responsible Party: Principal Investigator, Sean Savitz, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-22-1005
Record Dates: First submitted 2023-01-27; First posted 2023-02-21 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: telerehabilitation
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation (VAST 2) (Experimental)
  Interventions: Other: Telerehabilitation (VAST 2)

INTERVENTIONS:
Other: Telerehabilitation (VAST 2) — The telehealth platform will be available by a web secure link accessible on a home computer or loaded on user friendly tablets that are customized for the patient's impairments. Telerehabilitation services will include 2 out of 3 disciplines: Occupational Therapy, Speech Therapy, Physical Therapy. All therapy interventions will be delivered by licensed therapists and will be based on patients' specific impairments and goals. Therapy intervention will be provided 3x/wk. for each of 2 disciplines. The intervention will be going on for 4 weeks which will total to 24 sessions. Self-management support with trained health coach will be integrated into 1 therapy session each week. An additional individual 30 minute session will occur with the health coach each week.

SUMMARY:
The purpose of this study is to assess feasibility of a virtual rehabilitation program in stroke patients and to assess treatment effects, patient goal attainment with self-guided rehabilitation activities, barriers to and facilitators of telerehab, hospital readmission events, and social determinants of health

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by the subject or legally authorized representative.
* Diagnosed with hemorrhagic or ischemic stroke
* Pre-stroke mRS is less than 3
* Qualifying Stroke Event must be confirmed by CT or MRI
* Recommended to participate in self-guided or in-person rehabilitation activities by a physician or rehabilitation therapist
* Must have sufficient cognitive and language abilities to comprehend verbal commands and to carry out the study assessments
* Able to access the internet
* Mild-moderate impairments in motor or cognitive function

Exclusion Criteria:

* History of neurological or other disease resulting in significant functional impairment (e.g. Parkinson's disease, motor neuron disease, moderate dementia, arthritis, contractures or fixed anatomical abnormality).
* Subjects with a severe comorbid disorder that has reasonable likelihood of limiting survival to less than 6 months.
* Any other conditions that, in the opinion of the investigators, would preclude safe and/or effective participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
The experience of the participant measured by the participant experience surveys | end of study (about 10 weeks after baseline)
Number of participants that completed all scheduled visits. | end of study (about 10 weeks after baseline)

SECONDARY OUTCOMES:
Change in impact of stroke as assessed by the Stroke Impact Scale (SIS) | Baseline, end of intervention (about 5 weeks after baseline)
  This is a A 59 item questionnaire whereby subjects identify the impact of treatment on strength, hand function, mobility, activities of daily living, memory, communication, emotion, and handicap. Item responses are scored on a 5-point Likert-style scale. A score of 1 = an inability to complete the item and a score of 5 = no difficulty experienced at all. A standardized score ranging from 0 to 100 is calculated for all domains, with higher scores indicating a higher quality of life
Change in quality of life as assessed by the Short Form (SF-12)health questionnaire | Baseline, end of intervention (about 5 weeks after baseline)
  This is a health related quality of life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Change in cognitive impairment as assessed by the Montreal Cognitive Assessment (MoCA) | Baseline, end of intervention (about 5 weeks after baseline)
  Total score on the Montreal Cognitive Assessment (MoCA) range from 0 to 30, with a higher score indicating a better outcome.
Change in depression as assessed by the Patient Health Questionnaire (PHQ8) | Baseline, end of intervention (about 5 weeks after baseline)
  This is an 8 item questionnaire and each is scored from 0-24 a higher number indicating more depression
Change in disability as assessed by the Modified Rankin Scale (mRS) | Baseline, end of intervention (about 5 weeks after baseline)
  This scale is scored from 0(no symptoms at all) to 6 (dead), with a higher score being the worst outcome
Patient goal attainment with self-guided rehabilitation activities as assessed by the Goal Attainment Measure for Stroke (GAMS). | week 2
  This is a 4-point scale for multiple aspects of goal attainment Total scale scores range from high of 8 to a low of 0, with higher scores indicating goal attainment
Patient goal attainment with self-guided rehabilitation activities as assessed by the Goal Attainment Measure for Stroke (GAMS). | week 3
  This is a 4-point scale for multiple aspects of goal attainment Total scale scores range from high of 8 to a low of 0, with higher scores indicating goal attainment
Patient goal attainment with self-guided rehabilitation activities as assessed by the Goal Attainment Measure for Stroke (GAMS). | week 4
  This is a 4-point scale for multiple aspects of goal attainment Total scale scores range from high of 8 to a low of 0, with higher scores indicating goal attainment
Patient goal attainment with self-guided rehabilitation activities as assessed by the Goal Attainment Measure for Stroke (GAMS). | week 5
  This is a 4-point scale for multiple aspects of goal attainment Total scale scores range from high of 8 to a low of 0, with higher scores indicating goal attainment
Patient goal attainment with self-guided rehabilitation activities as assessed by the Goal Attainment Measure for Stroke (GAMS). | week 10
  This is a 4-point scale for multiple aspects of goal attainment Total scale scores range from high of 8 to a low of 0, with higher scores indicating goal attainment
Type of technology used by stroke patients as assessed by a questionnaire | end of intervention (about 5 weeks after baseline)
  Data will be reported categorically as number who use each type of technology, including cell phone, smart phone, tablet, laptop, and desktop.
Type of internet access used by stroke patients as assessed by a questionnaire | end of intervention (about 5 weeks after baseline)
  Data will be reported categorically as number who use each type of internet access including private wifi,public wifi, mobile data, hotspot, broadband
Use of computer equipment by stroke patients as assessed by a questionnaire | end of intervention (about 5 weeks after baseline)
  Data will be reported categorically as number who use each type of computer equipment , including a mouse and headphones
Type of issues exhibited when using the telehealth platform by stroke patients as as assessed by a questionnaire | end of intervention (about 5 weeks after baseline)
  Data will be reported categorically as number who face issues such as difficulty connecting to the telehealth platform, difficulty accessing/turning on camera, difficulty accessing/turning on audio and difficulty with calls being dropped
Number of stroke patients who exhibited any issues when they use the telehealth platform | end of intervention (about 5 weeks after baseline)
Type of technology used by caregivers as assessed by a questionnaire | end of intervention (about 5 weeks after baseline)
  Data will be reported categorically as number who use each type of technology, including cell phone, smart phone, tablet, laptop, and desktop.
Type of internet access used by caregivers as assessed by a questionnaire | end of intervention (about 5 weeks after baseline)
  Data will be reported categorically as number who use each type of internet access including private wifi,public wifi, mobile data, hotspot, broadband
Use of computer equipment by caregivers as assessed by a questionnaire | end of intervention (about 5 weeks after baseline)
  Data will be reported categorically as number who use each type of computer equipment , including a mouse and headphones
Type of issues exhibited when using the telehealth platform by caregivers as assessed by a questionnaire | end of intervention (about 5 weeks after baseline)
  Data will be reported categorically as number who face issues such as difficulty connecting to the telehealth platform, difficulty accessing/turning on camera, difficulty accessing/turning on audio and difficulty with calls being dropped
Number of caregivers who exhibited any issues when they use the telehealth platform | end of intervention (about 5 weeks after baseline)
Incidence of events that may lead to hospital readmission and falls as assessed by the adverse events | end of intervention (about 5 weeks after baseline)
Number of patients living in underserved areas | Baseline
Number of patients living in under resourced neighborhoods | Baseline
Socio Economic Status (SES) of patients as assessed by the patient demographics | Baseline
Housing condition of patients as assessed by the patient demographics | Baseline
Diastolic blood pressure assessed during virtual sessions using a web-based rehabilitation platform. | week 2
Diastolic blood pressure assessed during virtual sessions using a web-based rehabilitation platform. | week 3
Diastolic blood pressure assessed during virtual sessions using a web-based rehabilitation platform. | week 4
Diastolic blood pressure assessed during virtual sessions using a web-based rehabilitation platform. | week 5
Systolic blood pressure assessed during virtual sessions using a web-based rehabilitation platform. | week 2
Systolic blood pressure assessed during virtual sessions using a web-based rehabilitation platform. | week 3
Systolic blood pressure assessed during virtual sessions using a web-based rehabilitation platform. | week 4
Systolic blood pressure assessed during virtual sessions using a web-based rehabilitation platform. | week 5

CONTACTS AND LOCATIONS:
Overall Officials: Sean Savitz, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No